CLINICAL TRIAL: NCT00490685
Title: Randomized Continuation, Dose Escalation Trial of Sorafenib in Patients With Advanced HCC With Radiological Progression on Prior Sorafenib Treatment (Phase II Study)
Brief Title: Dose Escalation of Sorafenib in Patients With Advanced Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Armando Santoro, MD, Istituto Clinico Humanitas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2006-004; EUDRACT 2007-000758-30
Record Dates: First submitted 2007-06-22; First posted 2007-06-25 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2009-08

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sorafenib (BAY-43-9006)

SUMMARY:
The aim of the study is to evaluate, after radiological progression, efficacy in patients treated with Sorafenib at a dose of 600 mg bid compared to that in patients treated with best supportive care.

Primary efficacy objective is progression free survival from randomization.

ELIGIBILITY:
Inclusion Criteria:

Patients with advanced/inoperable HCC not eligible for radical or loco-regional therapies Male or female patients ≥ 18 years of age Life expectancy of at least 12 weeks at screening Histologically or cytologically documented HCC

At least one tumor lesion that meets both of the following criteria:

1. The lesion is measurable as per RECIST criteria, and
2. The lesion has not been subject to previous loco-regional therapy (such as radiation therapy, TACE, TAE, PEI, RFA, or cryoablation) Patients previously treated with loco-regional treatments are eligible provided that previously treated lesions are not selected as target lesions. Local therapy must be completed at least 4 weeks prior to the baseline scan ECOG PS of 0, 1, or 2 Cirrhotic status of Child-Pugh class A or B Barcelona-Clinic Liver Cancer (BCLC) stage B or C

The following laboratory parameters:

* Platelet count ≥ 60 x 109 /L
* Haemoglobin ≥ 8,5 g/dL
* Total bilirubin ≤ 3 mg/dL
* Alanine transaminase (ALT) and Aspartato transaminase (AST) ≤ 5 x upper limit of normal
* Amylase and lipase < 1,5 x the upper limit of normal
* Serum creatinine ≤ 1,5 x the upper limit of normal
* Prothrombin time (PT)-international normalized ratio (INR) < 2,3 or PT < 0,6 seconds above control. Patients who are being therapeutically anticoagulated with an agent such as Coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.

Written informed consent prior to any study specific screening procedures with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from HCC, except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1).
* Any cancer curatively treated > 3 years prior to entry is permitted Renal failure requiring hemo- or peritoneal dialysis
* History of cardiac disease: congestive heart failure > New York Heart Association (NYHA) class 2;
* active coronary artery disease (CAD);
* cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers ordigoxin), or uncontrolled hypertension.
* Myocardial infarction more than 6 months prior to study entry is permitted if there is no evidence of active CAD
* Active clinically serious infections (> Grade 2 [NCI CTCAE] )
* Known history of human immunodeficiency virus (HIV) infection
* Known Central Nervous System tumors including metastatic brain disease
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry
* History of organ allograft
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Patients unable to swallow oral medications
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study drug.
* Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy

REFERENCES:
- [Background] Abou-Alfa GK, Schwartz L, Ricci S, Amadori D, Santoro A, Figer A, De Greve J, Douillard JY, Lathia C, Schwartz B, Taylor I, Moscovici M, Saltz LB. Phase II study of sorafenib in patients with advanced hepatocellular carcinoma. J Clin Oncol. 2006 Sep 10;24(26):4293-300. doi: 10.1200/JCO.2005.01.3441. Epub 2006 Aug 14. PMID 16908937
- [Derived] Rimassa L, Pressiani T, Boni C, Carnaghi C, Rota Caremoli E, Fagiuoli S, Foa P, Salvagni S, Cortesi E, Chiara Tronconi M, Personeni N, Bozzarelli S, Chiara Banzi M, Fanello S, Romano Lutman F, Giordano L, Santoro A. A phase II randomized dose escalation trial of sorafenib in patients with advanced hepatocellular carcinoma. Oncologist. 2013;18(4):379-80. doi: 10.1634/theoncologist.2012-0221. Epub 2013 Apr 11. PMID 23580239